CLINICAL TRIAL: NCT02116244
Title: A Phase II, Open-label, Tolerability and Efficacy Study of Civamide Nasal Solution, 0.01%, in Patients With Dry Eye Syndrome
Brief Title: Civamide Nasal Solution for the Treatment of Dry Eye
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Winston Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WL-1001-08-02
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Dry Eye
Keywords: Dry Eye; Civamide; Zucapsaicin; Neuropeptides; TRPV-1
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Civamide Nasal Spray (Experimental): Civamide Nasal Spray 0.01% 20ug/dose (20ul), 10ul in each nostril, twice daily for 12 weeks
  Interventions: Drug: Civamide Nasal Spray

INTERVENTIONS:
Drug: Civamide Nasal Spray

SUMMARY:
Keratoconjunctivitis sicca (KCS) or Dry Eye Syndrome is a disease of the surface of the eye, tear film, and related ocular tissues. Millions of people suffer from one form of the disease or another and its prevalence increases with age. Dry Eye Syndrome sufferers experience a broad range of symptoms including discomfort, irritation, burning, itching, redness, pain, gritty feeling, foreign body sensation, blurred vision and ocular fatigue. Civamide is a TRPV-1 receptor modulator that causes the initial stimulation of neuropeptide release and subsequent desensitization to further stimulation of the trigeminovascular system. This provides a pharmacological rational for intranasal route of administration for disorders mediated by the trigeminal nerve or involving the cranial nerve. In nine clinical studies of Civamide Nasal Solution, over 50% of the nearly 300 patients who received Civamide via intranasal administration experienced lacrimation (tearing). This led to the hypothesis that Civamide Nasal Solution might be an appropriate treatment for Dry Eye Syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be aged 18 years or older.
2. Patients must have documented moderate to severe evaporative Dry Eye Syndrome for at least 6 months.
3. Patients must have a Schirmer (with anesthesia) of ≤ 8 per 5 minutes in at least one eye at Screening and Baseline (Day 1).
4. Patients must have a calculated overall score on the OSDI of >0.1 with no more than three responses of not applicable (N/A) at Screening and Baseline (Day 1).
5. Patients must have normal lid position and closure.
6. Women must be post-menopausal ≥ 1 year, or surgically sterilized. If not, a negative urine pregnancy test is required within 14 days of Day 1.
7. Informed consent must be provided.

Exclusion Criteria:

1. Patients with severe inflammatory Dry Eye Syndrome.
2. Patients with Dry Eye Syndrome secondary to Sjögren's Syndrome.
3. Patients with Schirmer (with anesthesia) of >8 per 5 minutes in both eyes.
4. Patients who are allergic to Civamide or any similar products, or excipients of Civamide Nasal Solution 0.01%.
5. Patients with history of previous ocular surgery or trauma.
6. Patients who require concurrent ocular medication for any eye disorder.
7. Patients who have used Restasis®, serum tears, or oral omega 3 supplements during the last 30 days or oral cyclosporine during the last 90 days.
8. Patients who are receiving or have received within 30 days any experimental systemic medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Schirmer Test | 12 Weeks
  Change in Schirmer Test from the Baseline Period to the last week (Week 12) of the Treatment Period.

SECONDARY OUTCOMES:
Schirmer Test | Week 1 and 6
  Change in Schirmer Test from the Baseline Period to the Score of each of weeks 1 and 6

OTHER OUTCOMES:
OSDI Patient Rating Assessment | Weeks 1, 6, and 12
  Change in the OSDI from the Baseline Period to Week 1, 6, and 12.
Investigator Rating Scale | Weeks 1, 6, and 12
  Investigator Rating Scale at Day 7, 42, and 84.
Requirement for Eye Lubricants | Weeks 1 to 12
  Requirement for Acute Medication

CONTACTS AND LOCATIONS:
Overall Officials: Scott B Phillips, MD, Study Director — Winston Laboratories
Locations (3):
- United States (3):
  - Wohl Eye Center, Bloomingdale, Illinois
  - NorthShore University HealthSystem, Glenview, Illinois
  - Chicago Cornea Consultants, Ltd., Hoffman Estates, Illinois

IPD SHARING:
Plan to Share IPD: No